CLINICAL TRIAL: NCT04140721
Title: Autonomic Determinants of Postural Tachycardia Syndrome (Chronic Pilot Study 2)
Brief Title: Autonomic Determinants of POTS - Pilot 2
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Andre' Diedrich, Research Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: VANDERBILT_IRB_191749; R01HL142583 (NIH)
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Postural Tachycardia Syndrome
Keywords: postural tachycardia syndrome; hyperadrenergic; moxonidine; sympatholytic; orthostatic symptoms; POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — moxonidine

STUDY DESIGN:
Intervention Model Description: randomized, double blind, crossover design
Who Masked: Participant, Investigator
Masking Description: Vanderbilt's Investigational Pharmacy will randomly assign participants to the moxonidine/placebo or placebo/moxonidine arm of the study. They will also provide the active drug and matching placebo. The medication distribution list will be kept by a dedicated person not involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moxonidine then Placebo (Experimental): After screening/baseline evaluations, patients will be discharged home on moxonidine 0.2-0.4 mg/day PO. After two weeks, the patients will be re-admitted for study testing while on moxonidine. At completion of this testing, patients will start taking matching placebo once daily PO to be continued at home. After two, the patients will be re-admitted for study testing while on placebo.
  Interventions: Drug: Placebo oral tablet; Drug: Moxonidine Pill
- Placebo then Moxonidine (Experimental): After screening/baseline evaluations, patients will be discharged home on placebo identical to moxonidine once daily PO. After two weeks, the patients will be re-admitted for study testing while on placebo. At completion of this testing, patients will start taking moxonidine 0.2-0.4 mg/day PO to be continued at home. After two weeks, the patients will be re-admitted for study testing while on moxonidine.
  Interventions: Drug: Placebo oral tablet; Drug: Moxonidine Pill

INTERVENTIONS:
Drug: Placebo oral tablet — Placebo pill identical to moxonidine administered for 4 weeks
  Other Names: inactive pill
Drug: Moxonidine Pill — Moxonidine pill administered for 4 weeks
  Other Names: Physiotens

SUMMARY:
Postural tachycardia syndrome (POTS) is a relatively common condition affecting mostly otherwise healthy young women. These patients have high heart rate and disabling symptoms during standing. Quality of life may be poor. The sympathetic nerves in the autonomic nervous system help to maintain normal blood pressures and heart rates during activities of daily life.

The purpose of this study is to determine the importance of sympathetic activation as a cause of orthostatic symptoms. The investigators will assess the effects of a blood pressure medication (Moxonidine) on the symptoms during standing. Moxonidine lowers sympathetic activity. The investigators believe patients with high resting sympathetic activity might benefit from Moxonidine. It might reduce high heart rate and improve symptoms during standing. This study should help clinicians and the growing population of patients with POTS gain a better understanding of this disorder and find more personalized treatment.

DETAILED DESCRIPTION:
Patients with POTS experience symptoms and an increase in heart rate≥30 beats/min with standing in the absence of orthostatic hypotension. As a result of considerable functional impairment, individuals with POTS are often unable to attend school or work. There is agreement that POTS is a heterogeneous disorder with multiple overlapping pathophysiologies proposed to underlie the clinical phenotype of patients. It would be important to define the underlying pathophysiological mechanisms in an individual patient to design optimal therapy. Our overarching hypothesis is that there is a subset of POTS patients (psPOTS) with a central sympathetic activation as the primary pathophysiology. We have characterized these patients by an increase in muscle sympathetic nerve activity (MSNA, a reflection of central sympathetic outflow) even at rest. In this project, we will focus on the role of primary sympathetic activation in the pathogenesis of POTS. Direct neural recordings of sympathetic activity, central sympathetic inhibition and extensive autonomic phenotyping will enable us to identify and correct the primary pathophysiology to optimally benefit psPOTS patients. This is a mechanistic study, designed to assess the effects of 4 weeks of central sympatholysis with moxonidine on orthostatic tachycardia and symptoms (Specific Aim 1), hypovolemia (Specific Aim 2) and central and peripheral baroreflex properties (Specific Aim 3) in a randomized, crossover design with POTS patients having elevated resting sympathetic nerve activity.

ELIGIBILITY:
Inclusion Criteria:

* meets criteria for postural tachycardia syndrome (POTS)

  1. a heart rate increase of ≥30 beats/min within 10 minutes of upright posture;
  2. lack of orthostatic hypotension (blood pressure fall ≥ 20/10 mmHg within 3 minutes of standing); and
  3. chronic symptoms during upright posture over at least 6 months, in the absence of any other acute cause.
* in the follicular phase of the menstrual cycle (days 5-13 of a 28-day cycle)
* POTS with primary central sympathetic activation (psPOTS) as defined as having resting MSNA ≥ 25 bursts/min
* able and willing to provide informed consent.

Exclusion Criteria:

* pregnancy,
* smoker,
* BMI>30 kg/m2,
* deconditioned status (if available VO2max<80% of predicted)
* unable to withdraw from medications known to affect autonomic function, blood pressure or blood volume
* systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathies, and autoimmune neuropathies.
* arteriosclerotic disease of carotid artery. History of neck surgery.
* conditions associated with inflammatory processes, such as coronary artery disease, hypertension, smoking, hypercholesterolemia (or on statin therapy), rheumatoid arthritis, diabetes,
* treatment with oral corticosteroids, current infections (e.g., urinary tract infection), or use of non-steroidal anti-inflammatory drugs.
* other factors which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Orthostatic Symptom Burden [delta (delta VOSS)] | after 30 min supine to after 15 min of 60 degrees upright tilt (delta VOSS), 2-3 hours after a dose of the treatment assigned for the previous period.
  VOSS is a validated questionnaire that consists of 9 items: mental clouding, blurred vision, shortness of breath, rapid heartbeat, tremulousness, chest discomfort, headache, lightheadedness, and nausea. Each item is scored on a 0 to 10 scale (with 0 reflecting absence of symptoms), and the change of the total scores (range: 0-90) from supine to upright postures (delta VOSS) will be used as a measure of orthostatic symptom burden. The primary outcome measure will be the difference in orthostatic symptom burden [delta (delta VOSS)] following 4 weeks of placebo vs. moxonidine treatment.

SECONDARY OUTCOMES:
Change in Orthostatic Change in Heart Rate [delta (delta HR)] | after 30 min supine to after 15 min of 60 degrees upright tilt (delta HR), 2-3 hours after a dose of the treatment assigned for the previous period.
  Difference in heart rate change from supine to upright postures (delta HR) following 4 weeks of placebo vs. moxonidine treatment [delta (delta HR)].

CONTACTS AND LOCATIONS:
Overall Officials: André Diedrich, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No